CLINICAL TRIAL: NCT04097535
Title: Determining the Magnitude of Early Steps of Fatty Acid Oxidation in Glioma Using 18F-FPIA
Brief Title: Measuring Fatty Acid Oxidation in Gliomas Using 18F-FPIA PET/MRI
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 18HH4394; 228245 (Other: IRAS)
Record Dates: First submitted 2019-09-17; First posted 2019-09-20 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-09

CONDITIONS: Glioma
Keywords: PET/MRI; Fatty Acid Oxidation
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Brain biopsy / surgical resection tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PET/MRI — Imaging scan

SUMMARY:
Glioma is the most common primary malignant brain tumour in adults and has an extremely poor prognosis. The aim of this study is to quantify the degree of early step fatty acid oxidation in gliomas as imaged by 18F-FPIA PET/MRI in 10 evaluable patients.

The Investigators hypothesise that FPIA uptake will be higher in high-grade gliomas compared to lower grade gliomas, in keeping with a higher propensity of high grade tumours to generate ATP and NADPH via fatty acid oxidation under bioenergetic stress.

DETAILED DESCRIPTION:
10 evaluable participants with suspected cerebral glioma on previous MRI who are due to undergo surgical resection or biopsy will be enrolled into the study. The patients invited to participate in the study will provide full consent, but will only undergo 18F-FPIA PET/MRI imaging once they have satisfied the inclusion and exclusion criteria. Once these have been satisfied, eligible participants will proceed to 18F-FPIA PET/MRI.

On the day of imaging the participants will undergo a blood test to measure plasma concentrations of carnitine. During the scan, a single dose of 18F-FPIA (maximum, 370 MBq) IV will be administered to the participant followed by a whole brain dynamic PET/MRI scan over 66 minutes. During the MRI sequences, the participant will receive an additional IV bolus of Gadolinium contrast medium administered through a peripheral venous cannula. Arterial blood sampling through a peripheral arterial line will be performed to determine the concentration of radiotracer within arterial plasma. All the participants that are enrolled into the study will undergo biopsy or surgical resection as part of their routine clinical care, from which their tumour grade will be confirmed; the Investigators will obtain tissue from these procedures to perform metabolomics, genomics and proteomics. Surgery or biopsy will be performed typically within 2 weeks but no later than 3 months.

ELIGIBILITY:
Inclusion Criteria:

Patients with radiological evidence of suspected cerebral glioma due for surgery or biopsy and with the following characteristics will be recruited:

* Age ≥18
* Tumour size at least 2 cm.
* WHO performance status 0 - 2.
* If female, the subject is either post-menopausal (at least 1 year), or surgically sterilized (has had a documented bilateral oophorectomy and/or documented hysterectomy for at least 2 years,), or if of childbearing potential, must have a negative urine beta human chorionic gonadotropin pregnancy test done at initial screening and on the day of tracer administration. The result of the pregnancy test must be known before administration of 18F-FPIA injection.
* The subject is able and willing to comply with study procedures, and signed and dated informed consent is obtained.
* The subject has a satisfactory medical history as judged by the investigator with no significant co-morbidities, physical examination, and vital signs findings during the screening period (from 21 days before administration).
* The subject's clinical and laboratory tests are within normal limits and/or considered clinically insignificant.

Exclusion

* The subject has received any chemotherapy, immunotherapy, biologic therapy or investigational therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of 18F-FPIA injection. The subject is pregnant or lactating.
* The subject is diabetic or has uncontrolled blood glucose or blood lipid levels (clinical decision by investigator), any other chronic illness that will preclude brief discontinuation of medication, or musculoskeletal condition that would not allow comfortable performance of a 66-minute study.
* The subject has received another investigational radioactive tracer within 1 month before administration of 18F-FPIA injection.
* Anticoagulation therapy, prolonged prothrombin time, abnormal Allen's test.
* Unsatisfactory renal function (eGFR<60)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with radiological evidence of suspected cerebral glioma due for surgery or biopsy
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Williams, MBChB, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Imperial College Healthcare NHS Trust/ Imperial College london, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Islam S, Inglese M, Grech-Sollars M, Aravind P, Dubash S, Barwick TD, O'Neill K, Wang J, Saleem A, O'Callaghan J, Anchini G, Williams M, Waldman A, Aboagye EO. Feasibility of [18F]fluoropivalate hybrid PET/MRI for imaging lower and higher grade glioma: a prospective first-in-patient pilot study. Eur J Nucl Med Mol Imaging. 2023 Nov;50(13):3982-3995. doi: 10.1007/s00259-023-06330-0. Epub 2023 Jul 25. PMID 37490079

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was open to recruitment from the 04Jun2018 to 07Aug2020.
  Intervention: [18F]FPIA injection and multi-parametric, multi-modal dynamic PET-MRI performed at Imanova Limited, Burlington Danes, Imperial College London (Hammersmith Hospital Campus), Du Cane Road, London, W12 0NN.
  The key objective of this study was to quantify the magnitude of the early steps fatty acid oxidation in human gliomas using [18F]FPIA PET/MRI.
Groups:
- Patients With a Suspected Cerebral Glioma on Standard of Care MRI: Participants with a suspected cerebral glioma on standard of care imaging that are enrolled into the study had an [18F]FPIA PET-MRI scan performed at Imanova Limited on a Signa™ 3.0 T scanner.
  All participants enrolled into the study subsequently underwent a biopsy or surgical resection as part of their routine clinical care. Tissue obtained post-procedure (surgical resection/biopsy) to determine tumour grade and perform metabolomics, genomics, and proteomics.
  PET-MRI Protocol: Subjects received a single I.V bolus injection of [18F]FPIA followed by a saline flush. A single dose of [18F]FPIA (maximum 370MBq) was administered followed by a whole brain dynamic PET-MRI scan over 66 minutes. During the MRI sequences, the patients received an additional I.V bolus of Gadolinium contrast-medium administered through a peripheral venous cannula.
  MRI: Sequences for attenuation correction of PET data (DIXON, zero-TE), volumetric T1-weighted images (pre- and post-contrast administration), volumetric T2, dynamic susceptibility contrast perfusion (DSC) and dynamic contrast enhanced perfusion (DCE).
  * Maximum Injected Activity: 370MBq
  * Conversion Factor (mSv/MBq): 0.0187
  * Total Effective Dose (mSv)/patient: 6.9 mSv
  The total effective dose for each patient in this study is 6.9 mSv. There is no ionising radiation from the MR component of the study.
Period: Overall Study
Arm/Group | Patients With a Suspected Cerebral Glioma on Standard of Care MRI
Started | 11
Completed | 10
Not Completed | 1
Not completed — [18F]FPIA/radiotracer production failure - Participant subsequently withdrew consent. | 1

BASELINE CHARACTERISTICS:
Groups:
- Patients With a Suspected Cerebral Glioma on Standard of Care MRI: Participants was a suspected cerebral glioma on standard of care imaging that are enrolled into the study had an [18F]FPIA PET-MRI scan performed at Imanova Limited on a Signa™ 3.0 T scanner.
  All participants enrolled into the study subsequently underwent a biopsy or surgical resection as part of their routine clinical care. Tissue obtained post-procedure (surgical resection/biopsy) to determine tumour grade and perform metabolomics, genomics, and proteomics.
  PET-MRI Protocol: Subjects received a single I.V bolus injection of [18F]FPIA followed by a saline flush. A single dose of [18F]FPIA (maximum 370MBq) was administered followed by a whole brain dynamic PET-MRI scan over 66 minutes. During the MRI sequences, the patients received an additional I.V bolus of Gadolinium contrast-medium administered through a peripheral venous cannula.
  MRI: Sequences for attenuation correction of PET data (DIXON, zero-TE), volumetric T1-weighted images (pre- and post-contrast administration), volumetric T2, dynamic susceptibility contrast perfusion (DSC) and dynamic contrast enhanced perfusion (DCE).
  * Maximum Injected Activity: 370MBq
  * Conversion Factor (mSv/MBq): 0.0187
  * Total Effective Dose (mSv)/patient: 6.9 mSv
  The total effective dose for each patient in this study is 6.9 mSv. There is no ionising radiation from the MR component of the study.
Arm/Group | Patients With a Suspected Cerebral Glioma on Standard of Care MRI
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 5
Age, Continuous [Mean (Full Range); unit: years] | 59.7 [31 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Quantitative Measurement of [18F]-FPIA Uptake in Human Gliomas
Description: Standardised uptake values (SUV) on [18F]FPIA PET/MRI
Time Frame: -21-0 days
Measure: Mean (Full Range); unit: SUV60_max
Groups:
- Patients With a Histologically Confirmed Grade II Glioma.: Participants with a suspected cerebral glioma on standard of care imaging that underwent an [18F]FPIA PET-MRI scan prior to routine biopsy/surgical resection. Tissue obtained post-procedure provided histological confirmation of a grade II glioma.
- Patients With a Histologically Confirmed Grade III Glioma.: Participants with a suspected cerebral glioma on standard of care imaging that underwent an [18F]FPIA PET-MRI scan prior to routine biopsy/surgical resection. Tissue obtained post-procedure provided histological confirmation of a grade III glioma.
- Patients With a Histologically Confirmed Grade IV Glioma.: Participants with a suspected cerebral glioma on standard of care imaging that underwent an [18F]FPIA PET-MRI scan prior to routine biopsy/surgical resection. Tissue obtained post-procedure provided histological confirmation of a grade IV glioma.
Arm/Group | Patients With a Histologically Confirmed Grade II Glioma. | Patients With a Histologically Confirmed Grade III Glioma. | Patients With a Histologically Confirmed Grade IV Glioma.
Number analyzed (Participants) | 2 | 3 | 5
SUV60_max | 0.9041 [0.8974 to 0.9108] | 1.3529 [1.1520 to 1.5910] | 2.0470 [1.6564 to 2.6358]

2. Secondary Outcome: Correlation of 18F-FPIA Uptake With Tumour Type and Histological Grade Including O6-methylguanine-DNA Methyltransferase (MGMT) and Isocitrate Dehydrogenase (IDH) Gene Expression.
Description: [18F]FPIA PET/MRI & Immunohistochemistry (IHC)
Time Frame: 0-3 months
Population: Five participants enrolled into the study were patients with a histologically confirmed grade IV glioma. IDH status and MGMT status were assessed separately using immunohistochemistry (IHC) for the five participants with a grade IV glioma.
Measure: Number; unit: participants
Arm/Group | Patients With a Histologically Confirmed Grade II Glioma. | Patients With a Histologically Confirmed Grade III Glioma. | Patients With a Histologically Confirmed Grade IV Glioma.
Number analyzed (Participants) | 2 | 3 | 5
participants
  IDH Status - IDH mutant | 2 | 3 | 0
  IDH Status - IDH wild-type | 0 | 0 | 5
  MGMT Status - MGMT Methylated: number analyzed (Participants) | 0 | 0 | 5
  MGMT Status - MGMT Methylated |  |  | 3
  MGMT Status - MGMT Unmethylated: number analyzed (Participants) | 0 | 0 | 5
  MGMT Status - MGMT Unmethylated |  |  | 2

ADVERSE EVENTS:
Time Frame: All adverse events were reported that had taken place up to 24 hours post injection of [18F]FPIA.
Arm/Group | Patients With a Suspected Cerebral Glioma on Standard of Care MRI
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT04097535/Prot_SAP_000.pdf